CLINICAL TRIAL: NCT00398606
Title: A Triple-Blind, Randomized, Active-Controlled, Parallel-Group, Multicenter Study to Evaluate and Compare the Efficacy and Tolerability of Alendronate Sodium With Calcium Supplementation in the Treatment of Osteoporosis in Postmenopausal Women
Brief Title: A Study to Compare the Efficacy of Alendronate With and Without Calcium or Calcium Alone In the Treatment of Osteoporosis in Postmenopausal Women (0217-088)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0217-088; 2006_546
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Alendronate; Duration of Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0217, alendronate sodium / Duration of Treatment : 2 Years
Drug: Comparator : calcium carbonate /Duration of Treatment : 2 Years

SUMMARY:
The purpose of this study is to see how well alendronate and calcium as compared to calcium alone increase bone density in postmenopausal women with osteoporosis

ELIGIBILITY:
Inclusion Criteria :

* Patient is postmenopausal (or surgically menopausal) for at least 5 years.
* Patient must be diagnosed with osteoporosis
* Patient has spinal anatomy suitable for DEXA of the lumbar spine

Exclusion Criteria :

* Patient is receiving or has received treatment prior to randomization which might influence bone turnover
* Patient has a history of or evidence for metabolic bone disease (other than postmenopausal bone loss)
* Patient is receiving or is expected to receive during the course of the study any medication (other than study medication) which might alter bone or calcium metabolism

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650
Dates: Start 1995-04; Primary Completion 1998-02 (Actual)

PRIMARY OUTCOMES:
BMD of the lumbar spine determined by a DEXA scan at 2 years

SECONDARY OUTCOMES:
BMD of the hip trochanter and femoral neck determined by a DEXA scan and biomarkers of bone turnover (BAP, NTX) at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Bonnick S, Broy S, Kaiser F, Teutsch C, Rosenberg E, DeLucca P, Melton M. Treatment with alendronate plus calcium, alendronate alone, or calcium alone for postmenopausal low bone mineral density. Curr Med Res Opin. 2007 Jun;23(6):1341-9. doi: 10.1185/030079907X188035. PMID 17594775